CLINICAL TRIAL: NCT06537102
Title: Unilateral Versus Bilateral Laparoscopic Ovarian Drilling In Clomiphene Citrate (CC) Resistant Cases of Polycystic Ovarian Syndrome (PCOS): A Randomized Controlled Study
Brief Title: Unilateral vs Bilateral Laparoscopic Ovarian Drilling In Clomiphene Citrate Resistant Cases of Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sahar Saeed Ahmed Elhalfawy, Resident of Obstetrics and Gynecology department, Ebiar central hospital, Faculty of Medicine, University of Tanta, Tanta, AL Gharbia ,, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34896/9/21
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Laparoscopic; Ovarian Drilling; Clomiphene Citrate; Polycystic Ovarian Syndrome; Unilateral; Bilateral
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral laparoscopic ovarian drilling group (Other): Patients underwent unilateral laparoscopic ovarian drilling Laparoscopic drilling was performed under general anesthesia as follows: 10-mm subumbilical entry and two 5-mm secondary ports in the lower part of the abdomen just above the anterior superior iliac spine. The laparoscope is introduced through the subumbilical port, and secondary ports was used for introduction of the instruments,the type of needle was an insulated unipolar needle electrode with a non-insulated distal end. We are planning to use the least thermal effective dose which is 60 J/cm3 of ovarian tissue.
  The number of punctures (Np) per ovary was calculated according to the following formula: N p = 60 J/cm3/40 W × 4 s, with 3 mm diameter and 4 mm depth for each puncture using power setting of 300 W for 2-4 s. Unilateral: was done on the larger ovary.
  Interventions: Other: Unilateral laparoscopic ovarian drilling
- Bilateral laparoscopic ovarian drilling group (Other): Laparoscopic drilling was performed under general anesthesia as follows: 10-mm subumbilical entry and two 5-mm secondary ports in the lower part of the abdomen just above the anterior superior iliac spine. The laparoscope is introduced through the subumbilical port, and secondary ports was used for introduction of the instruments,the type of needle was e an insulated unipolar needle electrode with a non-insulated distal end. We are planning to use the least thermal effective dose which is 60 J/cm3 of ovarian tissue.
  The number of punctures (Np) per ovary was calculated according to the following formula: N p = 60 J/cm3/40 W × 4 s, with 3 mm diameter and 4 mm depth for each puncture using power setting of 300 W for 2-4 s. Bilateral : using dose adjusted according to ovarian volume.
  Interventions: Other: Bilateral laparoscopic ovarian drilling

INTERVENTIONS:
Other: Unilateral laparoscopic ovarian drilling — Laparoscopic drilling was performed under general anesthesia as follows: 10-mm subumbilical entry and two 5-mm secondary ports in the lower part of the abdomen just above the anterior superior iliac spine. The laparoscope is introduced through the subumbilical port, and secondary ports was used for introduction of the instruments, the type of needle was an insulated unipolar needle electrode with a non-insulated distal end. We are planning to use the least thermal effective dose which is 60 J/cm3 of ovarian tissue.
  The number of punctures (Np) per ovary was calculated according to the following formula: N p = 60 J/cm3/40 W × 4 s, with 3 mm diameter and 4 mm depth for each puncture using power setting of 300 W for 2-4 s. Unilateral: was done on the larger ovary.
  Arms: Unilateral laparoscopic ovarian drilling group
Other: Bilateral laparoscopic ovarian drilling — Laparoscopic drilling was performed under general anesthesia as follows: 10-mm subumbilical entry and two 5-mm secondary ports in the lower part of the abdomen just above the anterior superior iliac spine. The laparoscope is introduced through the subumbilical port, and secondary ports was used for introduction of the instruments, the type of needle was an insulated unipolar needle electrode with a non-insulated distal end. We are planning to use the least thermal effective dose which is 60 J/cm3 of ovarian tissue.
  The number of punctures (Np) per ovary was calculated according to the following formula: N p = 60 J/cm3/40 W × 4 s, with 3 mm diameter and 4 mm depth for each puncture using power setting of 300 W for 2-4 s. Bilateral: Using dose adjusted according to ovarian volume.
  Arms: Bilateral laparoscopic ovarian drilling group

SUMMARY:
The aim of the current study is to compare the efficacy of laparoscopic unilateral ovarian drilling with bilateral ovarian drilling in clomiphene citrate resistant cases of polycystic ovarian syndrome in terms of clinical response (regularity of the cycle), change in biochemical parameters, ovulation rate over six months, pregnancy rate within six months.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS), is considered the most common endocrine disorder in reproductive age in females. Polycystic ovary syndrome (PCOS) is characterized by reproductive and metabolic disturbances. Androgen excess is a hallmark of polycystic ovary syndrome (PCOS), driving many of the phenotypic features

The clinical response to laparoscopic ovarian drilling (LOD) seems to be thermal energy dose-dependent. Two punctures (300 J) per ovary are associated with poor results. Between three and five (450-750 J) punctures per ovary seem to represent the effective thermal dose. The application of six or more (C900 J) punctures per ovary may result in excessive destruction to the ovary and should therefore be discouraged.

ELIGIBILITY:
Inclusion Criteria:

* Age within 25-35 years.
* Polycystic ovarian syndrome as diagnosed according to modified Rotterdam criteria 2018: oligomenorrhea or amenorrhea; clinical and/or biochemical signs of hyperandrogenism; and transvaginal sonographic appearance of polycystic ovaries (≥ 20 follicles or an ovarian volume 10 cm3) .
* Infertile women who have clomiphene citrate -resistant polycystic ovary syndrome (150 mg/daily for 5 days for six cycles with no ovulation).
* Normal semen analysis in the husband.

Exclusion Criteria:

* Hyper-androgenic disorders like late onset congenital adrenal hyperplasia, hyperprolactinemia, thyroid diseases.
* Cushing's syndrome and androgen-secreting tumors.
* Body mass index > 30 kg/m2.
* Other medical problems like diabetes, Hypertesion, patients on steroid hormone …. etc.
* Other causes of infertility as multiple uterine fibroids.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with Polycystic Ovarian Syndrome
Enrollment: 130 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Restoration of ovulation | 6 month after operation.
  Restoration of ovulation was measured before operation and for 6 month after operation .

SECONDARY OUTCOMES:
Folliculometry | 6 month after operation.
  Folliculometry was measured before operation and for 6 month after operation .
Follicle-stimulating hormone (FSH) | 6 month after operation.
  Follicle-stimulating hormone (FSH) was measured before operation and for 6 month after operation .
Luteinizing hormone (LH) | 6 month after operation.
  Luteinizing hormone (LH) was measured before operation and for 6 month after operation .
Anti-müllerian hormone(AMH) | 6 month after operation.
  Anti-müllerian hormone(AMH) was measured before operation and for 6 month after operation .
Pregnancy rate | 6 month after operation.
  Pregnancy rate was measured before operation and for 6 month after operation .

CONTACTS AND LOCATIONS:
Locations (1):
- Sahar Saeed Ahmed Elhalfawy, Tanta, ElGharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data was available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data was available upon a reasonable request from the corresponding author